CLINICAL TRIAL: NCT05614362
Title: The Effect of Channa Striatus Extract on Serum Albumin and High Sensitive C-Reactive Protein in End-Stage Renal Disease Patients
Brief Title: Channa Striatus Extract on Albumin and Hs-CRP ESRD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitas Sebelas Maret (Other)
Responsible Party: Principal Investigator, Nurhasan Agung Prabowo, Principal Investigator, Universitas Sebelas Maret
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CStriatusAlbHsCRP
Record Dates: First submitted 2022-10-20; First posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: End-Stage Renal Disease; Inflammation
Keywords: end-stage renal disease; albumin; hs-crp; randomized controlled trial; channa striatus
MeSH Terms: conditions — Kidney Failure, Chronic; Inflammation | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Channa striatus extract (Experimental): Channa striatus group was given 3x1 500mg dose of Channa striatus for 21 days
  Interventions: Dietary Supplement: Channa Striatus extract
- Placebo (Placebo Comparator): Placebo group was given 3x1 dose of maltodextrin for 21 days
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Channa Striatus extract — Channa Striatus extract given with a dose of 500 mg three-times-daily for each patient
  Arms: Channa striatus extract
Dietary Supplement: Maltodextrin — Maltodextrin given three-times-daily for each patient
  Arms: Placebo

SUMMARY:
This study is a randomised, double blind, placebo-controlled study in patients with ESRD on HD or CAPD based RRTs at Moewardi General Hospital in Surakarta, Indonesia from January to March 2021. Subjects were randomized to either a Channa striata or a placebo group and were given a three times daily dosage of 500 mg of Channa striatus extract or 500 mg maltodextrin, respectively for 21 days. Serum albumin and hs-CRP were measured at the baseline, and at the end of the study

DETAILED DESCRIPTION:
Study design This research was a randomized, double blinded, 2-arm parallel comparative study of CS extract vs placebo. This was conducted at the Department of Kidney and Hypertension, Moewardi General Hospital Surakarta from January 2021 - March 2021. The researcher has obtained an ethical clearance from the local ethics commission for basic/clinical research at Moewardi General Hospital, Surakarta.

Patient selection The population in this study were ESRD patients aged between 18 and 60 years old who underwent HD and CAPD at Moewardi General Hospital, Surakarta and agreed to being included in this study. Patients with history of malignancies, autoimmune disease, and active infection all were excluded. Patients who had taken any form albumin, herbal supplementation, antioxidant, steroid, immunosuppressive or heparin medication were also excluded. Sample selection was done by consecutive sampling to all eligible ESRD patients. The samples in this study would be divided into 2 groups; treatment group and control group, each had the same proportion of HD and CAPD patient.

Randomization and blinding The participants were randomized into 2 equal size groups which were the CS and placebo group. Participants were numbered sequentially following time of participation, and the type of RRT received. This separation of numbering according to RRT was performed to ensure an equal proportion of RRT received in both groups. A randomization list was generated using Random Allocation Software and subject numbers were allocated with 1:1 ratio, separately according to the type of RRT received. Blinding of participants and attending physicians were achieved by using identical capsules of placebo and CS extract.

The intervention The CS extract was obtained from ONOIWA® capsules (PT. Natura Nuswantara Nirmala, Tangerang, Indonesia) and purchased from a retail drug store. Each capsule contained pure 500 mg CS extract powder. The placebo used was 500 mg maltodextrin powder encapsulated in the same capsule color of the CS extract capsule. The placebo was prepared in Pharmacy Department of Moewardi General Hospital, and pre-purchased from a commercial drug store. Both of the groups consumed the extract of the placebo, with a dose of three times a day for 21 days.

Study visit and endpoint The venous blood samples for hs-CRP and albumin were collected before the administration of intervention, and at day 21. All of the tubes were then sent to the Department of Clinical Pathology at Moewardi General Hospital for the blood analysis to be performed. All social demographic feature of the patients were collected at baseline, including gender, age, type and length of RRT treatment. All of the patients were then monitored at each weekly visit to examine their clinical status and will be drop-outed when clinical deterioration occurred.

ELIGIBILITY:
Inclusion Criteria:

* ESRD patient
* Undergoing HD or CAPD

Exclusion Criteria:

* History of malignancy, autoimmune disease, active infection
* Supplementation of albumin, herbal, antioxidant, steroid, immunosuppresive, heparin

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Change of concentration of serum albumin | 21 days post-intervention
  Serum albumin is measured by laboratory assessment
Change of concentration of serum hs-CRP | 21 days post-intervention
  hs-CRP is measured by laboratory assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Moewardi General Hospital, Surakarta, Middle Java, Indonesia

IPD SHARING:
Plan to Share IPD: No